CLINICAL TRIAL: NCT00856388
Title: A Pilot Trial Of Reduced Intensity Allogeneic Stem Cell Transplantation With Fludarabine, Melphalan, And Low Dose Total Body Irradiation
Brief Title: Fludarabine Phosphate, Melphalan, Total-Body Irradiation, Donor Stem Cell Transplant in Treating Patients With Hematologic Cancer or Bone Marrow Failure Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 118807; NCI-2009-01508 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Aplastic Anemia; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Fanconi Anemia; Juvenile Myelomonocytic Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Paroxysmal Nocturnal Hemoglobinuria; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Anemia, Aplastic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, Large B-Cell, Diffuse; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Fanconi Anemia; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Hemoglobinuria, Paroxysmal; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — fludarabine phosphate; Melphalan; Whole-Body Irradiation; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Reduced intensity allogeneic stem cell transplant) (Experimental): Patients receive fludarabine phosphate IV over 30 minutes on days -5 to -2 and melphalan* IV over 30 minutes on day -2. Patients then undergo total-body irradiation on day -1 and allogeneic stem cell transplantation on day 0.
  Note: *Patients with chromosomal breakage syndromes, such as Fanconi anemia or dyskeratosis congenita, receive anti-thymocyte globulin IV over 4 hours on day -4 to -2 instead of melphalan.
  Interventions: Drug: fludarabine phosphate; Drug: melphalan; Radiation: total-body irradiation; Procedure: allogeneic hematopoietic stem cell transplantation; Biological: anti-thymocyte globulin

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Radiation: total-body irradiation — Undergo total-body irradiation
  Other Names: TBI
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic stem cell transplantation
Biological: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin

SUMMARY:
This clinical trial is studying how well giving fludarabine phosphate and melphalan together with total-body irradiation followed by donor stem cell transplant works in treating patients with hematologic cancer or bone marrow failure disorders. Giving low doses of chemotherapy and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells or abnormal cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer or abnormal cells (graft-versus-tumor effect)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the transplant related mortality (TRM) of this reduced intensity transplantation (RIT) combination in a patient population that is usually not eligible for a full myeloablative allogeneic transplant.

SECONDARY OBJECTIVES:

I. To evaluate engraftment, safety, clinical response, evidence of graft-versus-malignancy effect/graft-versus-host disease (GVHD) and overall outcomes of treatment with our RIT regimen across a variety of hematological conditions.

OUTLINE: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -5 to -2 and melphalan* IV over 30 minutes on day -2. Patients then undergo total-body irradiation on day -1 and allogeneic stem cell transplantation on day 0.

Note: *Patients with chromosomal breakage syndromes, such as Fanconi anemia or dyskeratosis congenita, receive anti-thymocyte globulin IV over 4 hours on day -4 to -2 instead of melphalan.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a histology documented hematologic malignancy or marrow disorder
* Bone marrow failure disorders and other non-malignant hematologic or immunologic disorders:

  * Acquired bone marrow failure disorders include aplastic anemia, paroxysmal nocturnal hemoglobinuria (PNH):

    * Primary allogeneic hematopoietic stem cell transplantation (HSCT) is appropriate for selected patients with severe aplastic anemia; however, patients with aplastic anemia must have failed at least one cycle of standard immunosuppressive therapy with calcineurin inhibitor plus anti-thymocyte globulin (ATG) if a fully-matched donor is not available
    * Patients with PNH must have a history of thrombosis related to PNH
  * Hereditary bone marrow failure disorders include Fanconi anemia or related chromosomal breakage syndrome dyskeratosis congenita, Diamond-Blackfan anemia, Shwachman-Diamond syndrome, Kostmann syndrome, congenital amegakaryocytic thrombocytopenia:

    * Fanconi anemia or related chromosomal breakage syndrome: positive chromosome breakage analysis using diepoxybutane (DEB) or mitomycin C if applicable
    * Dyskeratosis: diagnosis is supported by using either telomerase reverse transcriptase (TERC) gene mutation in autosomal dominant Dyskeratosis Congenita or Xlinked DKC1 gene mutation
  * Other non-malignant hematologic or immunologic disorders that require transplantation

    * Quantitative or qualitative congenital platelet disorders (including but not limited to congenital amegakaryocytopenia, absent-radii syndrome, Glanzmann's thrombasthenia)
    * Quantitative or qualitative congenital neutrophil disorders (including but not limited to chronic granulomatous disease, congenital neutropenia)
    * Congenital primary immunodeficiencies (including but not limited to Severe Combined Immunodeficiency Syndrome, Wiskott-Aldrick syndrome, CD40 ligand deficiency, T-cell deficiencies)
* Acute leukemias:

  * Subjects must be ineligible for conventional myeloablative transplantation;
  * Resistant or recurrent disease after at least one standard combination chemotherapy regime or first remission patients at high risk of relapse OR First remission patients at high risk of relapse:
  * Acute myeloid leukemia (AML)- antecedent myelodysplastic syndrome, secondary AML, high risk cytogenetic abnormalities or normal cytogenetics with high-risk molecular features (e.g. Flt3-ITD mutation, mixed-lineage leukemia [MLL], wildtype NPM1);
  * Acute lymphocytic leukemia (ALL)- high or standard risk ALL
* Chronic Myeloid Leukemia (CML):

  * Chronic phase (intolerant or unresponsive to imatinib and/or other tyrosine kinase inhibitors), second chronic phase or accelerated phase who are ineligible for conventional myeloablative transplantation
* Myeloproliferative and myelodysplastic syndromes (MDS):

  * Myelofibrosis (with/without splenectomy) with intermediate to high risk features
  * Advanced polycythemia vera not responding to standard therapy
  * MDS with an international prostate symptom score (IPSS) score of Int-2 or higher
  * MDS with lower IPSS scores Int-1 or less with severe clinical features such as severe neutropenia or thrombocytopenia or high risk chromosome abnormalities such as monosomy 7
  * Secondary massively parallel signature sequencing (MPSS) with any IPSS scores
  * Chronic myelomoncytic leukemia
* Lymphoproliferative disease:

  * Chronic lymphocytic leukemia (CLL), low-grade non-Hodgkin lymphoma (NHL) (recurrent or persistent) fludarabine refractory or with less than 6 months duration of complete response (CR) between courses of conventional therapy
  * Multiple myeloma, progressive disease after autologous stem cell transplant or as planned tandem (allogeneic transplant after prior autologous stem cell transplant)
  * Waldenstroms macroglobulinemia (failed one standard regimen)
  * High grade NHL and diffuse large B-cell lymphoma (DLBCL)
  * Not eligible for conventional myeloablative HSCT OR failed autologous HSCT
  * First remission lymphoblastic lymphoma, or small, non-cleaved cell lymphoma or mantle cell lymphoma
* Hodgkin disease:

  * Relapsed or refractory after front-line therapy
  * Failed or were not eligible for autologous transplantation
* Failed prior autotransplant
* Age >= 3 and =< 75 years for blood and bone marrow transplants and age >= 3, < 60 for cord blood transplants
* No serious uncontrolled psychiatric illness
* No concomitant active malignancy other than non-melanoma skin cancer
* Non-pregnant and non-nursing women (women or men with reproductive potential should agree to use an effective means of birth control)
* Patients may have received prior autologous bone marrow transplant (BMT) or prior myeloablative allogeneic BMT (at least 60 days have elapsed)
* At least 2 weeks since prior chemotherapy, radiation treatment and/or surgery
* Informed consent
* DONOR: Permissible HLA matching: Related donors- single antigen mismatch at HLA A, B or DRB 1; unrelated donors- a single antigen mismatch at HLA A, B, or C, +/- additional single allele level mismatch at A, B, C or DRB1; cord blood >= 4 out of 6 antigen match at HLA A, B, DRB1)
* DONOR: Compatibility at the four most informative HLA loci: A, B, C and DRB1 are important for reducing the risk of GVHD and successful transplant outcomes; the A, B, C and DRB1 loci comprise 8 possible alleles (a haplotype being inherited from each parent); one additional locus, HLA-DQ, is also typed to ascertain haplotypes and assist in the search for a compatible donor; however mismatching at DQ has not been shown to be associated with adverse outcomes; high resolution molecular typing (at the allele level) is now the standard of care for unrelated donor searches and allows greater refinement of the search strategy
* DONOR: Matched related donor: a single antigen mismatch at A, B, or the DR transplant from a family member is associated with a higher risk of GVHD but similar overall survival when compared to full identity at these 3 regions; related donor/recipient pairs must be matched at 5 of 6 HLA antigens (A, B, DRBl)
* DONOR: Unrelated donor: when evaluating patients for unrelated donor transplant, a higher degree of matching is preferred due to minimize the risk of GVHD; the A, B, C, DRB1 and DQ loci, comprising 10 possible alleles, will be typed routinely for all unrelated transplants; given the higher risk of TRM in mismatched transplants, RIT is often the best way to mitigate the risk; evolving data from the National Marrow Donor Program now makes it possible to estimate the risks of donor-recipient HLA mismatch at the allele or antigen level; the higher risk from HLA-mismatching must be carefully assessed with respect to the clinical urgency and the patient's risk by the transplant physician; antigen level mismatches at DQ are inconsequential to transplant outcomes and are ignored with respect to donor selection for the purposes of this protocol, with matching requirements confined to the 8 loci involving HLA A, B, C and DRB1; for the purpose of this protocol, a single antigen mismatch at HLA A, B, or C, with or without additional single allele level mismatch may participate in this protocol for voluntary unrelated donors (blood or marrow); patients must be at least antigen-level matched at DRB1
* DONOR: If a patient has no suitable family donor matched for 5 of 6 HLA antigens (A, B, DRB1) and no suitable unrelated donor is identified or for reasons of urgency, the patient can be considered a candidate for cord blood transplant, provided a cord blood donor is identified with a >= 4 out of 6 antigen match at HLA A, B, DRB1 antigens; the cord blood product must provide a minimum of 2 x 10^7 nucleated cells/kg, test negative for HIV and Hepatitis A, Band C, and sterility assays have no growth; the cord blood products are located through the National Marrow Donor Program, the American Registry, or the Bone Marrow Donor Worldwide or other established registries, and may be stored in the N.Y Placental Cord Blood Bank, the St. Louis Cord Blood Bank, or any of the established, registered International blood and marrow banks
* DONOR: Donor must be healthy and have nonreactive test results for all infectious disease assays as required by state and federal regulations; donors who screen seropositive for hepatitis and/or syphilis must be cleared by infectious disease consultation
* DONOR: The donor must have no uncontrolled cardiopulmonary, renal, endocrine, hepatic or psychiatric disease to render donation unsafe
* DONOR: The donor must be able to give informed consent for peripheral blood stem cell collection or bone marrow collection
* DONOR: Syngeneic donors are not eligible
* DONOR: Donors who have poor peripheral venous access, may require central venous line placement for stem cell apheresis

Exclusion Criteria:

* Uncontrolled central nervous system (CNS) disease (for hematologic malignancies)
* Karnofsky (adult) or Lansky (for =< 16 years) performance status =< 50%
* Diffusing capacity of the lung for carbon monoxide (DLCO) less than 40% predicted, corrected for hemoglobin (Hb) and/or alveolar ventilation
* Cardiac: left ventricular ejection fraction less than 40%
* Bilirubin >= 3 x upper limit of normal
* Liver alkaline phosphatase >= 3 x upper limit of normal
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvate transaminase (SGPT) >= 3 x upper limit of normal
* Child's class B and C liver failure
* Calculated creatinine clearance < 40 cc/min by the modified Cockcroft-Gault formula for adults or the Schwartz formula for pediatrics
* Patients who have received maximally allowed doses (given in 2 Gy fractions, or equivalent) of previous radiation therapy to various organs as follows:

  * Mediastinum 40 Gy
  * Heart (any volume) 36 Gy
  * Whole lungs 12 Gy
  * Small bowel (any volume) 46 Gy
  * Kidneys 12 Gy
  * Whole liver 20 Gy
  * Spinal cord (any volume) 36 Gy
  * Whole brain 30 Gy Enrollment of patients who previously receive higher than allowed dose of radiation to a small volume of lungs, liver, and brain will be determine by the discretion of the radiation oncologist on the study
* Uncontrolled diabetes mellitus, cardiovascular disease, active serious infection or other condition which, in the opinion of treating physician, would make this protocol unreasonably hazardous for the patient
* Human immunodeficiency virus (HIV) positive
* Patients who in the opinion of the treating physician are unlikely to comply with the restrictions of allogeneic stem cell transplantation based on formal psychosocial screening
* Females of childbearing potential with a positive pregnancy test

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-01-14 (Actual); Primary Completion 2012-08-09 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Chen, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Started | 62
Completed | 61
Not Completed | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 43
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Day 100 TRM
Description: Day 100 Treatment Related Mortality An exact 95% confidence interval will be provided.
Time Frame: First 100 days
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Number analyzed (Participants) | 61
percentage of participants | 8.44 [3.08 to 17.29]

2. Secondary Outcome: Median Time to ANC Engraftment
Description: Median Time to ANC Engraftment
  Summarized using standard descriptive statistics along with corresponding 95% confidence intervals.
Time Frame: Days 30
Population: All treated and eligible patients
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Number analyzed (Participants) | 61
Days | 16.5 [0 to 26]

3. Secondary Outcome: Median Time to Platelet Engraftment
Description: Median Time to Platelet Engraftment
  Summarized using standard descriptive statistics along with corresponding 95% confidence intervals.
Time Frame: Day 100
Population: All treated and eligible patients
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Number analyzed (Participants) | 61
Days | 17.0 [0 to 74]

4. Secondary Outcome: Rate of Complete Donor Chimerism - Blood
Description: Rate of Complete Donor Chimerism - Blood
  Summarized using standard descriptive statistics.
Time Frame: Day 30
Population: All treated and eligible patients, who were able to complete testing
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Number analyzed (Participants) | 44
percentage of participants | 89

5. Secondary Outcome: Rate of Complete Donor Chimerism - Blood
Description: Rate of Complete Donor Chimerism - Blood
  Summarized using standard descriptive statistics.
Time Frame: Day 100
Population: All treated and eligible patients, who were able to complete testing
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Number analyzed (Participants) | 49
percentage of participants | 94

6. Secondary Outcome: Acute GVHD Grade III-IV
Description: Acute GVHD grade III-IV
  Summarized using standard descriptive statistics along with corresponding 95% confidence intervals.
Time Frame: Up to day 100
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Number analyzed (Participants) | 61
percentage of participants | 27 [16 to 38]

7. Secondary Outcome: 1 yr Extenstive Chronic GVHD
Description: 1 yr Extensive Chronic GVHD
  Summarized using standard descriptive statistics along with corresponding 95% confidence intervals.
Time Frame: Up to 4.5 years
Population: All treated and eligible who survived to day 100 and were eligible to get chronic GVHD
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Number analyzed (Participants) | 53
percentage of participants | 60 [45 to 73]

8. Secondary Outcome: 3 yr Overall Survival
Description: 3 yr Overall Survival estimated using the Kaplan-Meier method.
Time Frame: Up to 4.5 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (Reduced Intensity Allogeneic Stem Cell Transplant): Patients receive fludarabine phosphate IV over 30 minutes on days -5 to -2 and melphalan* IV over 30 minutes on day -2. Patients then undergo total-body irradiation on day -1 and allogeneic stem cell transplantation on day 0.
  Note: *Patients with chromosomal breakage syndromes, such as Fanconi anemia or dyskeratosis congenita, receive anti-thymocyte globulin IV over 4 hours on day -4 to -2 instead of melphalan.
  fludarabine phosphate: Given IV
  melphalan: Given IV
  total-body irradiation: Undergo total-body irradiation
  allogeneic hematopoietic stem cell transplantation: Undergo allogeneic stem cell transplantation
  anti-thymocyte globulin: Given IV
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Number analyzed (Participants) | 61
percentage of participants | 46.0 [33.0 to 57.0]

ADVERSE EVENTS:
Arm/Group | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant)
Serious Adverse Events (participants affected / at risk) | 34/62
Other Adverse Events (participants affected / at risk) | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Reduced Intensity Allogeneic Stem Cell Transplant) (N=62)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (3)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 5 (5)
Disease progression (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (6)
Graft versus host disease (Immune system disorders) | 8 (9)
Bacteraemia (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (3)
Renal failure (Renal and urinary disorders) | 2 (3)
Urinary tract disorder (Renal and urinary disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 12 (16)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes